CLINICAL TRIAL: NCT06952855
Title: Observational Study to Evaluate Effectiveness, Safety and Satisfaction Level of Zastaprazan (JAQBO®) Under Daily Treatment for Patients With Erosive Gastroesophageal Reflux Disease
Brief Title: Observationa Study is a Prospective and Multi-institutional Observational Study.
Status: Completed | Type: Observational
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: JL-JAQ-401
Record Dates: First submitted 2025-03-11; First posted 2025-05-01 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Erosive Reflux Disease; Heartburn; Acid Regurgitation
Keywords: GERD; ERD
MeSH Terms: conditions — Heartburn; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 1 cohort: No interventions

SUMMARY:
This observational study is a prospective, multi-institutional non intervention study to examine the prescription patterns, corresponding treatment effects and safety in routine clinical practice for patients prescribed for the treatment of gastroesophageal reflux disease.

DETAILED DESCRIPTION:
The present observational study is designed to check effect and safety for patients who have been prescribed JAQBO for the treatment of erosive gastroesophageal reflux disease.

ELIGIBILITY:
Inclusion Criteria:

1. An adult over 19 years of age
2. A person who voluntarily provides written informed consent

Exclusion Criteria:

1. A pregnant woman or a nursing woman
2. A person who is deemed unsuitable for the subject of the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: GERD patients
Sampling Method: Non-Probability Sample
Enrollment: 5536 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Change in GERD (heartburn, acid regurgitation) score in RDQ | 4 weeks
  Scale(none / 1day / 2day/ 3-4 day / 5-6 day/ every day)

CONTACTS AND LOCATIONS:
Locations (1):
- Goodbreath Medical Center, Seoul, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided